CLINICAL TRIAL: NCT07206147
Title: Physical Exercise as Treatment Post-stroke Fatigue - a Feasibilty Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other); Strokeförbundet (Unknown); Hjärnskadefonden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 282165
Record Dates: First submitted 2025-07-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Fatigue Symptom
Keywords: Post-stroke fatigue; Stroke; Physical exercise; Physical activity; Physiotherapy
MeSH Terms: conditions — Stroke; Fatigue; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FaStEx (Experimental)
  Interventions: Other: FaStEx - Structured strength training
- Control group (Active Comparator)
  Interventions: Other: Control group

INTERVENTIONS:
Other: FaStEx - Structured strength training — Strength training in group session, 2 times a week for 8 weeks. 150 minutes of physical activity per week that is carried out independently.
  Arms: FaStEx
Other: Control group — 150 minutes of physical activity per week that is carried out independently.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility the treatment FaStEx (FatigueStrokeExercise) which consists of strength exercise in people with brain fatigue after stroke, referred to as post-stroke fatigue. The main questions it aims to answer are:

* What is the feasibility of a study with the treatment FaStEx, structured physical training, for people with post-stroke fatigue?
* What factors are important for people with post-stroke fatigue to be able to complete the FaStEx treatment?
* How do people with post-stroke fatigue experience participation in the study with the FaStEx treatment?

Researchers will compare FaStEx to physical activity at home to see if FaStEx can reduce post-stroke fatigue.

Participants will

* Carry out strength training twice a week at a health care center.
* Carry out physical activity for at least 150 minutes per week on their own. Participants in the control group will carry out this physical activity as well.
* The treatment lasts for eight weeks.

DETAILED DESCRIPTION:
Type of treatment FaStEx (FatigueStrokeExercise) - Structured physiotherapist-led exercise intervention.

Dose Strength training for 45 minutes, twice a week for eight weeks.

Components of exercises All training sessions will have the same structure and consist of warm-up, strength training and cool-down.

Each training session starts with a 10-minute warm-up on an exercise bike or through body movements. The strength training is performed as station training with one participant/station. The stations consist of eight different exercises. The participant performs 12 repetitions, 3 sets/exercise, 30 seconds rest between each set. Then rest and transfer to the next station, about 1 min. The load should be 10-12 RM and as a load are used body weight, dumbbells, gym machines, rubber bands, weight cuffs or kettlebells.

Exercises

1. Legs - leg press, squat or raise.
2. Arms - biceps curls (dumbbells or rubber bands).
3. Legs - Knee extension with load (gym machine, weight cuff, rubber band, cable station).
4. Shoulder - lat pull down (gym machine, rubber band).
5. Core - sit-ups or other core training.
6. Shoulder - rowing (cable station, rubber bands, dumbbells).
7. Balance - stand on one leg, tandem standing.
8. Legs - step-up board.

The training session ends with a cool-down through body movements and stretching.

Estimation of exertion with Borg RPE and brain fatigue with VAS before and after the session.

Place The training sessions are carried out in a training room at a health center.

Modifications Alternative exercises will be suggested by the instructor if necessary, e.g. the need for other equipment or support during the exercise. Participants are encouraged to perform the exercises to the best of their ability.

Choice of instructor The instructors are licensed physiotherapists who work in primary care in Region Örebro County who are used to instructing and individualizing training.

Home training In addition to the structured physiotherapist-led training, all participants in the study (control and intervention group) should independently perform aerobic physical activity of at least 150 min/v at a moderate intensity (Borg RPE 12-13). In connection with the start of the intervention, the participants receive an advisory conversation about physical activity to support how they can achieve 150 min/week.

Adherence Participation in strength training will be noted by the treating physiotherapist. Adherence to achieving physical activity for 150 min/w will be followed by participants filling out an activity diary.

ELIGIBILITY:
Inclusion Criteria:

- Stroke ≥6 months, able to move independently ≥100 meters with or without a walking aid, speak Swedish, Fatigue assessment scale (FAS) ≥24 points

Exclusion Criteria:

* Other neurological disease. Severe impairment of vision, hearing and/or cognition that prevents participation in the intervention. Already performs structured strength training (e.g. gym, group training) regularly (at least 1 time/week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue assessment scale | Baseline. End of treament at 8 weeks.
  Change in fatigue. 10-item Numerical Self-Rating Scale. Each item of the FAS is answered using a five-point, Likert-type scale ranging from 1 ("never") to 5 ("always"). Items 4 and 10 are reverse-scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.

SECONDARY OUTCOMES:
Chair stand test. | Baseline. End of treament at 8 weeks.
  Change in leg strength. Records the number of stands a person can complete in 30 seconds.
Activities-specific Balance Confidence Scale | Baseline. End of treament at 8 weeks.
  Change in confidence in one's balance ability. 16-item Numerical Self-Rating Scale. Each item is answered using a scale ranging from 0 % ("No confidence") to 100 % ("Completely confident"). Total scores can range from 0, indicating the lowest level of confidence, to 100 , denoting the highest.
Patient health questionnaire | Baseline. End of treament at 8 weeks.
  Change in depression. 9-item Numerical Self-Rating Scale. Each item is answered using a three-point, Likert-type scale ranging from "0" (not at all) to "3" (nearly every day). Total scores can range from 0, indicating no depression, to 27, denoting severe depression.
6 minute walking test | Baseline. End of treament at 8 weeks.
  Change in aerobic capacity and walking ability. The test subject walks back and forth over a measured distance of 30 m at a self-selected speed. The test measures pulse, blood pressure, self-estimated exertion and distance walked.
RAND 36 | Baseline. End of treament at 8 weeks.
  Change in quality of life. 36-item Numerical Self-Rating Scale with multiple choice options. Total scores can range from 0, indicating worse quality of life, to 100, denoting better quality of life.
Levels of physical activity | Measurement will take place 1 week before baseline and 1 week after the intervention at 8 weeks.
  Measured with accelerometer. The accelerometer is a small device worn on the thigh that measures movement in three planes.
Sedentary time | Measurement will take place 1 week before baseline and 1 week after the intervention at 8 weeks.
  Measured with accelerometer. The accelerometer is a small device worn on the thigh that measures movement in three planes.
Levels of physical activity (self-reported) | Measurement will take place continuously from baseline to end of treatment at 8 weeks
  Assessed with activity diary. The participants make notes of their physical activity during the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Örebro county, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No